CLINICAL TRIAL: NCT00003933
Title: The Incidence and Prognostic Significance of P16 INK4A/ P15 INK4B Gene Alterations in Children With Relapsed ALL Treated on CCG-1941
Brief Title: Diagnostic Study of Gene Alterations in Children Who Have Been Treated for Relapsed Acute Lymphocytic Leukemia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Purpose: Diagnostic
Other Study IDs: B9805; COG-B9805 (Other: Children's Oncology Group); CCG-B9805 (Other: Children's Cancer Group); CDR0000067125 (Other: Clinical Trials.gov)
Record Dates: First submitted 1999-11-01; First posted 2003-05-02 (Estimated); Last update posted 2014-08-07 (Estimated); Status verified 2014-08

CONDITIONS: Leukemia
Keywords: recurrent childhood acute lymphoblastic leukemia
MeSH Terms: conditions — Leukemia; Precursor Cell Lymphoblastic Leukemia-Lymphoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: laboratory biomarker analysis

SUMMARY:
RATIONALE: Diagnostic procedures, such as genetic testing, may improve the ability to detect acute lymphocytic leukemia and determine the extent of disease.

PURPOSE: Diagnostic study to try to detect changes in the genes of children who have been treated for relapsed acute lymphocytic leukemia.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the incidence of p16/p15 homozygous deletions and p15 promoter hypermethylation in acute lymphocytic leukemia cells of children treated on protocol CCG-1941.
* Determine the prognostic importance of p16/p15 abnormalities in these children.
* Determine the presence or absence of p16/p15 abnormalities in the dominant clone at diagnosis if present at relapse in these patients.

OUTLINE: Frozen cells are obtained from samples collected on protocol CCG-1941. DNA is isolated and examined using Southern blot analysis to assay for deletions and promoter hypermethylation of p16 and/or p15.

PROJECTED ACCRUAL: Approximately 100 samples will be obtained for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of acute lymphocytic leukemia and treated on protocol CCG-1941
* Material cryopreserved in the CCG cell bank

PATIENT CHARACTERISTICS:

Age:

* Children

Performance status:

* Not specified

Life expectancy:

* Not specified

Hematopoietic:

* Not specified

Hepatic:

* Not specified

Renal:

* Not specified

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* Not specified

Chemotherapy:

* Not specified

Endocrine therapy:

* Not specified

Radiotherapy:

* Not specified

Surgery:

* Not specified

Other:

* See Disease Characteristics

Max Age: 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Dates: Start 1999-04; Primary Completion 2006-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stephen P. Hunger, MD, Study Chair — University of Florida
Locations (41):
- United States (38):
  - Long Beach Memorial Medical Center, Long Beach, California
  - Children's Hospital Los Angeles, Los Angeles, California
  - Jonsson Comprehensive Cancer Center, UCLA, Los Angeles, California
  - Children's Hospital of Orange County, Orange, California
  - UCSF Cancer Center and Cancer Research Institute, San Francisco, California
  - David Grant Medical Center, Travis Air Force Base, California
  - Children's Hospital of Denver, Denver, Colorado
  - Children's National Medical Center, Washington D.C., District of Columbia
  - Shands Hospital and Clinics, University of Florida, Gainesville, Florida
  - University of Chicago Cancer Research Center, Chicago, Illinois
  - Indiana University Cancer Center, Indianapolis, Indiana
  - Holden Comprehensive Cancer Center, Iowa City, Iowa
  - University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan
  - CCOP - Kalamazoo, Kalamazoo, Michigan
  - University of Minnesota Cancer Center, Minneapolis, Minnesota
  - Mayo Clinic Cancer Center, Rochester, Minnesota
  - Children's Mercy Hospital, Kansas City, Missouri
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Saint Peter's University Hospital, New Brunswick, New Jersey
  - Cancer Institute of New Jersey, New Brunswick, New Jersey
  - NYU School of Medicine's Kaplan Comprehensive Cancer Center, New York, New York
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - Mount Sinai School of Medicine, New York, New York
  - Herbert Irving Comprehensive Cancer Center, New York, New York
  - Lineberger Comprehensive Cancer Center, UNC, Chapel Hill, North Carolina
  - Veterans Affairs Medical Center - Fargo, Fargo, North Dakota
  - CCOP - Merit Care Hospital, Fargo, North Dakota
  - Children's Hospital Medical Center - Cincinnati, Cincinnati, Ohio
  - Ireland Cancer Center, Cleveland, Ohio
  - Children's Hospital of Columbus, Columbus, Ohio
  - Doernbecher Children's Hospital, Portland, Oregon
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Children's Hospital of Pittsburgh, Pittsburgh, Pennsylvania
  - Vanderbilt-Ingram Cancer Center, Nashville, Tennessee
  - University of Texas - MD Anderson Cancer Center, Houston, Texas
  - Children's Hospital and Regional Medical Center - Seattle, Seattle, Washington
  - Fred Hutchinson Cancer Research Center, Seattle, Washington
  - University of Wisconsin Comprehensive Cancer Center, Madison, Wisconsin
- Princess Margaret Hospital for Children, Perth, Western Australia, Australia
- Canada (2):
  - British Columbia Children's Hospital, Vancouver, British Columbia
  - IWK Health Centre, Halifax, Nova Scotia